CLINICAL TRIAL: NCT04768738
Title: The Effect Of Transcutaneous Auricular Vagus Nerve Stimulation On Sports Performance And Physiological Parameters In Healthy Young Individuals: Randomized, Double-Blind Study
Brief Title: The Effect Of Transcutaneous Auricular Vagus Nerve Stimulation On Sports Performance And Physiological Parameters
Acronym: VNS001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Principal Investigator, SEFA HAKTAN HATIK, PT, MSc, PhD(c), Sinop University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: VNS001
Record Dates: First submitted 2021-02-03; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy; Activity, Motor
Keywords: Transcutaneous auricular Vagus Nerve Stimulation; Sportive Performance; Physiological Parameters
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 46 healthy young individuals aged 19.2±1.5 years participated in the study. The participants were randomly divided into 3 groups as Above Threshold Group (n:15; 10 females, 5 males), Under Threshold Group (n:15; 10 females, 5 males) and Control Group (no stimulation) (n:16; 11 females, 5 males) according to the sensation of electrical current on ears. The participants were evaluated 3 times; before the application, after the first and second bicycle exercises. Numerical pain scale (NPS), pulse rate, blood pressure, respiratory rate, and distance travelled during exercise for sportive performance were recorded in kilometers as the evaluation method. The stimulation was done during the first bicycle exercise with 5 minutes of duration. The Kruskal-wallis, mann-whitney u test were used for the quantitative independent data obtained. In the analysis of qualitative independent data, chi-squared test was used.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Above Threshold Group (Experimental): In the above threshold group, biphasic current was applied as follows; frequency 10 Hz, in Modulation mode (Modulation mode is a combination of pulse rate and pulse width modulation. The pulse rate and width are automatically varied in a cycle pattern. The pulse width is reduced by 50% from its original setting in 0.5 second, then the pulse rate is reduced by 50% from its original setting in 0.5 second. Total cycle time is 1 second.), the pulse width was 300 μs. The current intensity was kept constant where the participant felt the current comfortably and applied for 5 minutes.
  Interventions: Device: Auricular Vagus Nerve Stimulation Level Of Above Threshold; Diagnostic Test: 5 Minutes Bicycle Exercise
- Subthreshold Group (Experimental): In the subthreshold group, biphasic current was applied as follows; frequency 10 Hz, in Modulation mode (Modulation mode is a combination of pulse rate and pulse width modulation. The pulse rate and width are automatically varied in a cycle pattern. The pulse width is reduced by 50% from its original setting in 0.5 second, then the pulse rate is reduced by 50% from its original setting in 0.5 second. Total cycle time is 1 second.), the pulse width was 300 μs. The parameters were the same with Above Threshold Group but the current was reduced to where the participant did not feel the current after the threshold value was reached and again applied for 5 minutes.
  Interventions: Device: Auricular Vagus Nerve Stimulation Level Of Subthreshold; Diagnostic Test: 5 Minutes Bicycle Exercise
- Control Group (Sham Comparator): In the control group, bicycle exercise was performed under the same load with the current-free headset produced for sham applications for 5 minutes. Participants were shown that the device was working, but no current was given.
  Interventions: Device: Auricular Vagus Nerve Stimulation Sham Method; Diagnostic Test: 5 Minutes Bicycle Exercise

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation Level Of Above Threshold — Biphasic current was applied as follows; frequency 10 Hz, in Modulation mode (Modulation mode is a combination of pulse rate and pulse width modulation. The pulse rate and width are automatically varied in a cycle pattern. The pulse width is reduced by 50% from its original setting in 0.5 second, then the pulse rate is reduced by 50% from its original setting in 0.5 second. Total cycle time is 1 second.), the pulse width was 300 μs. The current intensity was kept constant where the participant felt the current comfortably and applied for 5 minutes.
  Arms: Above Threshold Group
Device: Auricular Vagus Nerve Stimulation Level Of Subthreshold — biphasic current was applied as follows; frequency 10 Hz, in Modulation mode (Modulation mode is a combination of pulse rate and pulse width modulation. The pulse rate and width are automatically varied in a cycle pattern. The pulse width is reduced by 50% from its original setting in 0.5 second, then the pulse rate is reduced by 50% from its original setting in 0.5 second. Total cycle time is 1 second.), the pulse width was 300 μs. The parameters were the same with Above Threshold Group but the current was reduced to where the participant did not feel the current after the threshold value was reached and again applied for 5 minutes.
  Other Names: Level Of Subthreshold
  Arms: Subthreshold Group
Device: Auricular Vagus Nerve Stimulation Sham Method — Participants were shown that the device was working, but no current was given.
  Other Names: Sham Method
  Arms: Control Group
Diagnostic Test: 5 Minutes Bicycle Exercise — Participants in this group were asked to perform bicycle exercise with maximum performance under 50 watts for 5 minutes.
  Other Names: Bicycle Exercise

SUMMARY:
OBJECTIVE: The aim of this study is to investigate the effect of non-invasive auricular VNS (Vagus Nerve Stimulation) on sportive performance and physiological parameters in healthy individuals.

MATERIAL AND METHOD: 46 healthy young individuals aged 19.2(±1.5) years participated in the study. The participants were randomly divided into 3 groups as Above Threshold Group (n:15; 10 females, 5 males), Under Threshold Group (n:15; 10 females, 5 males) and Control Group (no stimulation) (n:16; 11 females, 5 males) according to the sensation of electrical current on ears. The participants were evaluated 3 times; before the application, after the first and second bicycle exercises. Numerical pain scale (NPS), pulse rate, blood pressure, respiratory rate, and distance travelled during exercise for sportive performance were recorded in kilometers as the evaluation method. The stimulation was done during the first bicycle exercise with 5 minutes of duration. The Kruskal-wallis, mann-whitney u test were used for the quantitative independent data obtained. In the analysis of qualitative independent data, chi-squared test was used.

DETAILED DESCRIPTION:
This study included 46 individuals aged 18-35 years in the home patient care laboratory at Sinop University Vocational School of Turkeli. Priorities were explained and the permission of the individuals was obtained. The number of females and males was divided into 3 groups as randomized. Participants were evaluated by Numerical pain scale (NPS), pulse rate, blood pressure, respiratory rate, and saturation measurement. In addition, the distance travelled during the exercise for sportive performance was recorded in kilometers. In the study, evaluation was conducted 3 times before the application, after the first and second bicycle exercises.

The study was double-blind randomized. Participants in the whole group were asked to perform bicycle exercise with maximum performance under 50 watts for 5 minutes. In all groups Vagustim device was used for stimulation. In the above threshold group, biphasic current was applied as follows; frequency 10 Hz, in Modulation mode (Modulation mode is a combination of pulse rate and pulse width modulation. The pulse rate and width are automatically varied in a cycle pattern. The pulse width is reduced by 50% from its original setting in 0.5 second, then the pulse rate is reduced by 50% from its original setting in 0.5 second. Total cycle time is 1 second.), the pulse width was 300 μs. The current intensity was kept constant where the participant felt the current comfortably and applied for 5 minutes. VNS was applied bilaterally to transmit current from the tragus and concha parts of the ear. After the first bicycle exercise, the participants were re-evaluated. In the second bicycle exercise, it was asked to perform for 5 minutes under the same load without any application. The study was evaluated for the third time and the study was completed.

In the subthreshold group, the parameters were the same but the current was reduced to where the participant did not feel the current after the threshold value was reached and again applied for 5 minutes. It was re-evaluated after the first bicycle exercise. In the second bicycle exercise, he was asked to perform bicycle exercise with maximum performance for 5 minutes under the same load without any application. The study was evaluated for the third time and the study was completed.

In the control group, bicycle exercise was performed under the same load with the current-free headset produced for sham applications for 5 minutes. Participants were shown that the device was working, but no current was given. It was re-evaluated after the first bicycle exercise. In the second bicycle exercise, the device was removed and asked to perform bicycle exercise with maximum performance for 5 minutes under the same load. The study was evaluated for the third time and the study was completed.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years age
* Being healthy

Exclusion Criteria:

* any known disease
* any drug usage

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Sportive performance | Change from Baseline at Second Exercise
  Athletic performance during exercise in healthy individuals, cycling length in kilometers. Measured twice, during first and second exercises.

SECONDARY OUTCOMES:
Pulse | Change from Baseline at 5 minutes
  Heart beats per minute. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Pulse | 15 minutes
  Heart beats per minute. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Numerical pain scale (NPS), | Change from Baseline at 15 minutes
  Amount of pain described by patients. Patients are asked to circle the number between 0 and 10. Zero represents 'no pain at all' whereas ten represents 'the worst pain ever possible'. Measurement is done twice; after the first and the second bicycle exercises.
Respiratory Rate | Change from Baseline at 5 minutes
  The respiratory rate corresponds to the number of breaths taken per minute. The rate of respiration measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Respiratory Rate | 15 minutes
  The respiratory rate corresponds to the number of breaths taken per minute. The rate of respiration measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Systolic Blood Pressure | Change from Baseline at 5 minutes
  Systolic Pressure measured 3 times; before the first exercise, after the first exercise, after the second exercise. Blood pressure recorded as mmHg. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Systolic Blood Pressure | 15 minutes
  Systolic Pressure measured 3 times; before the first exercise, after the first exercise, after the second exercise. Blood pressure recorded as mmHg. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Diastolic Blood Pressure | Change from Baseline at 5 minutes
  Diastolic Pressure measured 3 times; before the first exercise, after the first exercise, after the second exercise. Blood pressure recorded as mmHg. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Diastolic Blood Pressure | 15 minutes
  Diastolic Pressure measured 3 times; before the first exercise, after the first exercise, after the second exercise. Blood pressure recorded as mmHg. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Saturation | Change from Baseline at 5 minutes
  Percentage of Oxygen saturation in blood. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.
Saturation | 15 minutes
  Percentage of Oxygen saturation in blood. Measured 3 times; before the first exercise, after the first exercise, after the second exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Sefa Haktan Hatık, Sinop, Turkeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nur Gökçe, E , Pınar Cengi̇z, Z , Erbaş, O . (2018). Uzun ömrün sırrı: Vagus siniri . İstanbul Bilim Üniversitesi Florence Nightingale Tıp Dergisi , 4 (3) , 154-165 . Retrieved from https://dergipark.org.tr/tr/pub/ibufntd/issue/39718/470405
- [Background] Tracey, K.J., Inhibition of inflammatory cytokine production by cholinergic agonists and vagus nerve stimulation. 2003, Google Patents
- [Background] Hong GS, Zillekens A, Schneiker B, Pantelis D, de Jonge WJ, Schaefer N, Kalff JC, Wehner S. Non-invasive transcutaneous auricular vagus nerve stimulation prevents postoperative ileus and endotoxemia in mice. Neurogastroenterol Motil. 2019 Mar;31(3):e13501. doi: 10.1111/nmo.13501. Epub 2018 Nov 8. PMID 30406957
- [Background] Liu JJ, Huang N, Lu Y, Zhao M, Yu XJ, Yang Y, Yang YH, Zang WJ. Improving vagal activity ameliorates cardiac fibrosis induced by angiotensin II: in vivo and in vitro. Sci Rep. 2015 Nov 24;5:17108. doi: 10.1038/srep17108. PMID 26596640
- [Background] Lataro RM, Silva CA, Fazan R Jr, Rossi MA, Prado CM, Godinho RO, Salgado HC. Increase in parasympathetic tone by pyridostigmine prevents ventricular dysfunction during the onset of heart failure. Am J Physiol Regul Integr Comp Physiol. 2013 Oct 15;305(8):R908-16. doi: 10.1152/ajpregu.00102.2013. Epub 2013 Aug 15. PMID 23948774
- [Background] Dalli J, Colas RA, Arnardottir H, Serhan CN. Vagal Regulation of Group 3 Innate Lymphoid Cells and the Immunoresolvent PCTR1 Controls Infection Resolution. Immunity. 2017 Jan 17;46(1):92-105. doi: 10.1016/j.immuni.2016.12.009. Epub 2017 Jan 5. PMID 28065837
- [Background] Penry JK, Dean JC. Prevention of intractable partial seizures by intermittent vagal stimulation in humans: preliminary results. Epilepsia. 1990;31 Suppl 2:S40-3. doi: 10.1111/j.1528-1157.1990.tb05848.x. PMID 2121469
- [Background] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part II. Headache. 2016 Feb;56(2):259-66. doi: 10.1111/head.12650. Epub 2015 Sep 18. PMID 26381725
- [Background] Straube A, Ellrich J, Eren O, Blum B, Ruscheweyh R. Treatment of chronic migraine with transcutaneous stimulation of the auricular branch of the vagal nerve (auricular t-VNS): a randomized, monocentric clinical trial. J Headache Pain. 2015;16:543. doi: 10.1186/s10194-015-0543-3. Epub 2015 Jul 9. PMID 26156114
- [Background] Silberstein SD, Calhoun AH, Lipton RB, Grosberg BM, Cady RK, Dorlas S, Simmons KA, Mullin C, Liebler EJ, Goadsby PJ, Saper JR; EVENT Study Group. Chronic migraine headache prevention with noninvasive vagus nerve stimulation: The EVENT study. Neurology. 2016 Aug 2;87(5):529-38. doi: 10.1212/WNL.0000000000002918. Epub 2016 Jul 13. PMID 27412146
- [Background] Tassorelli C, Grazzi L, de Tommaso M, Pierangeli G, Martelletti P, Rainero I, Dorlas S, Geppetti P, Ambrosini A, Sarchielli P, Liebler E, Barbanti P; PRESTO Study Group. Noninvasive vagus nerve stimulation as acute therapy for migraine: The randomized PRESTO study. Neurology. 2018 Jul 24;91(4):e364-e373. doi: 10.1212/WNL.0000000000005857. Epub 2018 Jun 15. PMID 29907608
- [Background] Beh SC, Friedman DI. Acute vestibular migraine treatment with noninvasive vagus nerve stimulation. Neurology. 2019 Oct 29;93(18):e1715-e1719. doi: 10.1212/WNL.0000000000008388. Epub 2019 Sep 25. PMID 31554650
- [Background] Busch V, Zeman F, Heckel A, Menne F, Ellrich J, Eichhammer P. The effect of transcutaneous vagus nerve stimulation on pain perception--an experimental study. Brain Stimul. 2013 Mar;6(2):202-9. doi: 10.1016/j.brs.2012.04.006. Epub 2012 May 7. PMID 22621941
- [Background] Moller M, Mehnert J, Schroeder CF, May A. Noninvasive vagus nerve stimulation and the trigeminal autonomic reflex: An fMRI study. Neurology. 2020 Mar 10;94(10):e1085-e1093. doi: 10.1212/WNL.0000000000008865. Epub 2020 Feb 6. PMID 32029547
- [Background] Colzato LS, Ritter SM, Steenbergen L. Transcutaneous vagus nerve stimulation (tVNS) enhances divergent thinking. Neuropsychologia. 2018 Mar;111:72-76. doi: 10.1016/j.neuropsychologia.2018.01.003. Epub 2018 Jan 8. PMID 29326067
- [Background] Oshinsky ML, Murphy AL, Hekierski H Jr, Cooper M, Simon BJ. Noninvasive vagus nerve stimulation as treatment for trigeminal allodynia. Pain. 2014 May;155(5):1037-1042. doi: 10.1016/j.pain.2014.02.009. Epub 2014 Feb 14. PMID 24530613
- [Background] Antonino D, Teixeira AL, Maia-Lopes PM, Souza MC, Sabino-Carvalho JL, Murray AR, Deuchars J, Vianna LC. Non-invasive vagus nerve stimulation acutely improves spontaneous cardiac baroreflex sensitivity in healthy young men: A randomized placebo-controlled trial. Brain Stimul. 2017 Sep-Oct;10(5):875-881. doi: 10.1016/j.brs.2017.05.006. Epub 2017 May 19. PMID 28566194
- [Background] Sabino-Carvalho, J.L., et al., Non-invasive Vagus Nerve Stimulation Acutely Improves Blood Pressure Control in a Placebo Controlled Study. The FASEB Journal, 2017. 31(1_supplement): p. 848.8-848.8.
- [Background] Annoni EM, Xie X, Lee SW, Libbus I, KenKnight BH, Osborn JW, Tolkacheva EG. Intermittent electrical stimulation of the right cervical vagus nerve in salt-sensitive hypertensive rats: effects on blood pressure, arrhythmias, and ventricular electrophysiology. Physiol Rep. 2015 Aug;3(8):e12476. doi: 10.14814/phy2.12476. PMID 26265746
- [Background] Tiedt N, Religa A. Vagal control of coronary blood flow in dogs. Basic Res Cardiol. 1979 May-Jun;74(3):266-76. doi: 10.1007/BF01907744. PMID 475732
- [Background] Chen M, Yu L, Liu Q, Jiang H, Zhou S. Vagus nerve stimulation: A spear role or a shield role in atrial fibrillation? Int J Cardiol. 2015 Nov 1;198:115-6. doi: 10.1016/j.ijcard.2015.06.171. Epub 2015 Jul 5. No abstract available. PMID 26184434
- [Background] Lee SW, Li Q, Libbus I, Xie X, KenKnight BH, Garry MG, Tolkacheva EG. Chronic cyclic vagus nerve stimulation has beneficial electrophysiological effects on healthy hearts in the absence of autonomic imbalance. Physiol Rep. 2016 May;4(9):e12786. doi: 10.14814/phy2.12786. PMID 27173672
- [Background] Annoni EM, Van Helden D, Guo Y, Levac B, Libbus I, KenKnight BH, Osborn JW, Tolkacheva EG. Chronic Low-Level Vagus Nerve Stimulation Improves Long-Term Survival in Salt-Sensitive Hypertensive Rats. Front Physiol. 2019 Jan 31;10:25. doi: 10.3389/fphys.2019.00025. eCollection 2019. PMID 30766489
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Yoo PB, Liu H, Hincapie JG, Ruble SB, Hamann JJ, Grill WM. Modulation of heart rate by temporally patterned vagus nerve stimulation in the anesthetized dog. Physiol Rep. 2016 Feb;4(2):e12689. doi: 10.14814/phy2.12689. PMID 26811057
- [Background] Xie X, Lee SW, Johnson C, Ippolito J, KenKnight BH, Tolkacheva EG. Intermittent vagal nerve stimulation alters the electrophysiological properties of atrium in the myocardial infarction rat model. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1575-8. doi: 10.1109/EMBC.2014.6943904. PMID 25570272
- [Background] Li M, Zheng C, Sato T, Kawada T, Sugimachi M, Sunagawa K. Vagal nerve stimulation markedly improves long-term survival after chronic heart failure in rats. Circulation. 2004 Jan 6;109(1):120-4. doi: 10.1161/01.CIR.0000105721.71640.DA. Epub 2003 Dec 8. PMID 14662714